CLINICAL TRIAL: NCT01119755
Title: Seasonal Variation of 24hour Ambulatory Blood Pressure Monitoring in Treated Hypertensives
Brief Title: Seasonal Variation of Ambulatory Blood Pressure
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George S. Stergiou, Professor of Medicine, University of Athens
Other Study IDs: SV
Record Dates: First submitted 2010-04-21; First posted 2010-05-10 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2011-12

CONDITIONS: Hypertension
Keywords: TREATMENT OF HYPERTENSION
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective study to evaluate the change in 24 hour ambulatory blood pressure during winter and summer in well controlled treated hypertensives.

DETAILED DESCRIPTION:
Two 24hour ambulatory blood pressure monitorings, 4 to 6 months apart, will be performed on hypertensive subjects on a stable antihypertensive drug therapy for at least 4 weeks.

The correlation of weather and temperature with the 24hour ambulatory blood pressure monitoring will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 yrs
* Treated hypertension on stable treatment for at least 8 weeks
* Average home blood pressure (at least 5 days, 20 readings) < 130/80 mmHg

Exclusion Criteria:

* Congestive heart failure
* Use of loop diuretics

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TREATED HYPERTENSIVES REFERRED TO AN OUTPATIENT CLINIC
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George S Stergiou, MD, Study Chair — Hypertension Center,Third Department of Medicine,University of Athens,Greece
Locations (1):
- Hypertension Center, Third Department of Medicine, University of Athens, Greece, Athens, Greece

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 49
Region of Enrollment [Number; unit: participants]
  Greece | 80

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference of Systolic Daytime Ambulatory Blood Pressure Between Summer and Winter.
Description: Mean difference of systolic daytime ambulatory blood pressure measurement during summer and winter period
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1
Number analyzed (Participants) | 80
mmHg | 7.7 (14)

2. Secondary Outcome: Mean Difference of Systolic Clinic Blood Pressure Between Summer and Winter
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1
Number analyzed (Participants) | 80
mmHg | 7.5 (11.1)

3. Primary Outcome: Mean Difference of Diastolic Daytime Ambulatory Blood Pressure Between Summer and Winter
Description: Mean Difference of Diastolic Daytime Ambulatory Blood Pressure Measurement During Summer and Winter Period
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1
Number analyzed (Participants) | 80
mmHg | 4.1 (10)

4. Primary Outcome: Mean Difference of Systolic Night-time Ambulatory Blood Pressure Between Summer and Winter
Description: Mean difference of systolic night-time ambulatory blood pressure measurement during summer and winter period
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1
Number analyzed (Participants) | 80
mmHg | -0.1 (11.2)

5. Primary Outcome: Mean Difference of Diastolic Night-time Ambulatory Blood Pressure Between Summer and Winter
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1
Number analyzed (Participants) | 80
mmHg | 0.6 (8.9)

6. Secondary Outcome: Mean Difference of Diastolic Clinic Blood Pressure Between Summer and Winter
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1
Number analyzed (Participants) | 80
mmHg | 2.7 (7)

7. Secondary Outcome: Mean Difference of Systolic Home Blood Pressure Between Summer and Winter
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1
Number analyzed (Participants) | 80
mmHg | 3.2 (14)

8. Secondary Outcome: Mean Difference of Diastolic Home Blood Pressure Between Summer and Winter
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1
Number analyzed (Participants) | 80
mmHg | 2.7 (4.1)

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes